CLINICAL TRIAL: NCT03755570
Title: How is COGNItive Function Affected by Cardiac Resynchronisation Therapy?
Acronym: COGNI-CRT
Status: Suspended | Type: Observational
Why Stopped: PI request
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 251230
Record Dates: First submitted 2018-11-21; First posted 2018-11-28 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Cognitive Impairment; Cognitive Change; Heart Failure, Systolic; Heart Failure; Cognitive Impairment, Mild; Left Ventricular Dysfunction; Left Ventricular Systolic Dysfunction; Systolic Dysfunction; Systolic Heart Failure
Keywords: Cognitive Impairment; Left Ventricular Systolic Dysfunction; Heart Failure; Cardiac Resynchronisation Therapy; Implantable Cardioverter-Defibrillator; Pacemaker; CRT; ICD; PPM
MeSH Terms: conditions — Cognitive Dysfunction; Heart Failure, Systolic; Heart Failure; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- CRT: Main Arm: Cardiac Resynchronisation Therapy (CRT): Main Arm ~98 participants
  Prior to CRT Implantation & Post-Implant 6-Month Device Follow-Up Clinic:
  - Battery of 5 questionnaire-based cognitive tests, including the Test of Premorbid Functioning, Repeatable Battery for the Assessment of Neuropsychological Status, Hospital Anxiety and Depression Scale, Frontal Assessment Battery and Trail Making Test Part A and B
  Please note, the Test of Premorbid Functioning will only be performed ONCE at Pre-Assessment as results reflect IQ prior to disease onset.
  Interventions: Diagnostic Test: Repeatable Assessment of Neuropsychological Status; Diagnostic Test: Hospital Anxiety and Depression Scale; Diagnostic Test: Frontal Assessment Battery; Diagnostic Test: Trail Making Test Part A and B; Diagnostic Test: Test of Premorbid Functioning
- ICD and PPM: Control Arm: Implantable Cardioverter-Defibrillator (ICD) and Permanent Pacemaker (PPM): Control Arm ~98 participants
  Prior to ICD or PPM Implantation & Post-Implant 6-Month Device Follow-Up Clinic:
  - Battery of 5 questionnaire-based cognitive tests, including the Test of Premorbid Functioning Repeatable Battery for the Assessment of Neuropsychological Status, Hospital Anxiety and Depression Scale, Frontal Assessment Battery and Trail Making Test Part A and B
  Please note, the Test of Premorbid Functioning will only be performed ONCE at Pre-Assessment as results reflect IQ prior to disease onset.
  Interventions: Diagnostic Test: Repeatable Assessment of Neuropsychological Status; Diagnostic Test: Hospital Anxiety and Depression Scale; Diagnostic Test: Frontal Assessment Battery; Diagnostic Test: Trail Making Test Part A and B; Diagnostic Test: Test of Premorbid Functioning

INTERVENTIONS:
Diagnostic Test: Repeatable Assessment of Neuropsychological Status — Cognitive Function Test (Questionnaire-based)
  Other Names: RBANS; Repeatable Battery for Assessment Neuropsychological Status
Diagnostic Test: Hospital Anxiety and Depression Scale — Cognitive Function Test (Questionnaire-based)
  Other Names: HADS
Diagnostic Test: Frontal Assessment Battery — Cognitive Function Test (Questionnaire-based)
  Other Names: FAB
Diagnostic Test: Trail Making Test Part A and B — Cognitive Function Test (Questionnaire-based)
  Other Names: TMT
Diagnostic Test: Test of Premorbid Functioning — Cognitive Function Test (Questionnaire-based)
  Other Names: TOPF

SUMMARY:
The primary objective of COGNI-CRT is to assess whether Cardiac Resynchronisation Therapy (CRT) can improve cognitive function in patients with systolic HF (LVEF ≤35%), when compared to a control group of patients implanted with an Implantable Cardioverter-Defibrillator (ICD) or a permanent pacemaker (PPM) with systolic HF (LVEF ≤35%).

This clinical investigation is a prospective, single-centre cohort study. Each participant will be followed for 6 months. The study will collect data over 3 years; 2.5 years for enrolment and 6 months until the last participant completes the last 6-month follow-up visit.

N.B: COGNI-CRT does NOT affect the patient's care pathway - the patients who will be selected for participation are those who have already been referred for the device implant. The ONLY difference to the patient's care pathway caused by COGNI-CRT is the addition of a battery of cognitive function tests, which involves asking the patient questions and asking them to complete questionnaire-like cognitive tests.

NTpro-BNP levels, NYHA classification and LVEF will be measured prior to device implantation and at 6-months post-implant to assess the device's impact on the participant's heart failure (and CRT response). N.B: NT-proBNP, NYHA classification and LVEF are all parts of the patient's standard care pathway, COGNI-CRT is just utilising the data collected as part of the investigation.

The main study arm and control group allows COGNI-CRT to assess 3 potential outcomes for patients with severe HF (LVEF <35%):

1. Cognitive function is not improved by CRT, ICDs or PPMs
2. Cognitive function can be improved by the assurance of rate control offered by CRT, ICDs and PPMs
3. Cognitive function can be improved by the assurance of ventricular synchronisation and rate control provided by the additional left ventricular lead in CRT devices.

DETAILED DESCRIPTION:
Purpose:

The purpose of this clinical investigation is to assess whether cardiac resynchronisation therapy (CRT) can improve cognitive function in patients with systolic heart failure (Left Ventricular Ejection Fraction (LVEF) ≤35%), when compared to a control group of patients implanted with an implantable cardioverter-defibrillator (ICD) or permanent pacemaker (PPM) with systolic heart failure (LVEF ≤35%).

Design:

This clinical investigation is a prospective, single-centre cohort study. The study will be conducted at the Royal Cornwall Hospital Trust (RCHT) in Cornwall, England. Subjects will be followed for 6 months.

Cognitive performance will be assessed in patients pre- and post-CRT implant (Group A). An ICD and PPM control group (Group B) will also be assessed using the same battery of cognitive function tests to ensure any difference in cognitive function which is identified between pre- and post- CRT implant is due to the CRT therapy, and not due to a placebo effect (which can be especially powerful with implanted devices) or due to a learning effect (i.e. patients tested on the second occasion might improve their scores because they have had more practice).

N.B: COGNI-CRT does NOT affect the patient's care pathway - the patients who will be selected for participation are those who have already been referred for the device implant. The ONLY difference to the patient's care pathway caused by COGNI-CRT is the addition of a battery of cognitive function tests, which involves asking the patient questions and asking them to complete questionnaire-like cognitive tests.

LVEF, NT-proBNP and New York Heart Association (NYHA) classification data which is collected prior to device implantation and at 6-months post-implant will be utilised for analysis to measure response to CRT and to assess difference between the main arm and control group.

Arms in the study will be:

* Group A: Participants implanted with a CRT who are eligible according to the inclusion/ exclusion criteria
* Group B: Participants implanted with an ICD or a PPM who are eligible according to the inclusion / exclusion criteria

Objectives:

Primary objective: To assess whether CRT can improve cognitive function in patients with systolic heart failure (LVEF ≤35%), when compared to a control group of patients implanted with an ICD or PPM with systolic heart failure (LVEF ≤35%).

Secondary Objectives:

* To assess whether CRT can improve cognitive function
* To assess whether ICD and PPM therapy can improve cognitive function
* To assess if the level of improvement in cognitive function correlates to LVEF improvement / stability and/or NYHA improvement /stability and/or NT-proBNP level reduction (CRT response).

Subject Population:

The subject population enrolled in this investigation will comprise of male and female patients aged 20-89 years old. These subjects are patients who are willing to provide informed consent and meet the specific eligibility criteria. A minimum of 198 participants will be enrolled in this investigation.

Data for this study will be collected at:

* Enrolment
* Pre-Assessment for CRT, ICD or PPM Implantation
* Cardiac Implantable Electronic Device (CIED) Implant
* Post-Implant 6-Week Device Check (For device optimisation)
* Post-Implant 6-Month Device Follow-Up Visit After completing the Post-Implant 6-Month Device Follow-Up Visit, the patient will have completed his/her participation in the study.

Devices Used:

Implanted CRT-P, CRT-D, ICD and PPM devices may include Biotronik, Boston Scientific, Medtronic and St Jude Medical.

Patient Screening:

Patients who are referred to RCHT for CRT, ICD or PPM implantation with systolic heart failure (LVEF ≤35%) will be screened prior to Pre-Assessment by the clinical team. Prospective patients will be afforded sufficient time to consider participation in COGNI-CRT.

Cognitive Tests Used to Evaluate Cognitive Function:

To be Performed Only At Pre-Assessment:

1. Test of Premorbid Functioning (TOPF): TOPF provides the participant with a list of 70 words that have atypical grapheme to phoneme translations. The participant must attempt to read the list aloud so pronunciation of the words can be assessed. This tests IQ and memory as the participant must be familiar with the words, rather than being able to spell out a word they do not know. It takes approximately 10 minutes to complete

   To be Performed at Pre-Assessment and at the Post-Implant 6-Month Device Follow-Up Visit:
2. Hospital Anxiety and Depression Scale (HADS): The test consists of 14 multiple-choice questions, each attempting to ascertain about the frequency the participant has felt a certain symptom within the last 7 days. There are 4 answers to choose from which range from suffering from the symptom "nearly all the time" to "not at all" and are graded 0-3 depending on the participant's answer.
3. Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): Consisting of 12 sections, to evaluate 5 types of cognitive function: immediate memory; visuospatial/ constructional; attention; language and delayed memory.
4. Frontal Assessment Battery (FAB): The test has 6 neuropsychological tasks which involve asking the participant questions, for example "In what way are a banana and an orange alike?", and learning simple actions in response to hand taps or movements.
5. Trail Making Test (TMT) Parts A & B: Both parts of TMT involve circles dotted over a piece of paper, the circles for Part A are marked with the numbers 1 - 25 and the patient must draw a line connecting the numbers in ascending order, i.e. "1-2-3-4-5-6…" etc. Part B involves numbers and letters dotted around the page, from 1-13 and from A-L. The patient must connect the numbers and letters in ascending order, alternating between numbers and letters, i.e. "1-A-2-B-3-C…" etc

Response to CRT Measures will be measured prior to device implantation and at the 6-month follow-up device follow-up clinic:

LVEF: LVEF will be measured prior to device implant to assess the patient's heart function, and at the Post-Implant 6-Month Device Follow-Up Visit.

NT-proBNP: NT-proBNP levels from the patient's routine blood tests prior to device implantation and at the Post-Implant 6-Month Device Follow-Up Visit where blood testing is routine for heart failure patients every 6 months.

NYHA: A NYHA scale assessment will be performed during the screening clinics prior to device implant, and at the Post-Implant 6-Month Device Follow-Up Visit using the standardised NYHA questions designed for the purpose of this trial.

N.B: The above 3 tests (LVEF, NT-proBNP and NYHA classification) are performed routinely as part of the patient standard care pathway for heart failure, and this data will be utilised for analysis in this trial. The tests are NOT performed for the purpose of COGNI-CRT.

Device Optimisation:

At the post-implant 6-week device follow-up check, all efforts will be made to ensure the device is optimised as much as is possible, and the patient listed for MDT if problems are encountered to attempt to resolve problems.

Data Analysis:

Data will be tested for normality. Tests for group differences will be used to compare cognitive function between patients before and after CRT implant, and in the control group before and after ICD or PPM implant. Tests for group differences will also be used in comparison of the LVEF values, BNP results, NYHA classification, QRS duration, percentage biventricular pacing and BP measurements. Sample size calculations have estimated the required CRT sample size to power the study to be 99 participants (with a 95% confidence interval and a 5% margin of error). The expectation is for 99 patients to sign the informed consent and complete follow-up = 99 CRT participants. The control group will aim to enrol a similar figure to the main study group, a further 99 ICD and PPM participants. 99 CRT patients + 99 ICD or PPM patients = 198 patients are expected to be enrolled and complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing implant of a CRT system with an LVEF of ≤35% (main group), or ICD or PPM system with an LVEF of ≤35% (control group)
* Are 20 - 89 years of age
* Be able to provide written informed consent prior to investigational related procedure, and be willing and able to comply with the described protocols and follow-up schedules listed in the PIS
* Be literate to a level in which the cognitive function tests can be completed effectively
* Mental capacity to provide informed consent and undertake cognitive function tests
* Geographically stable and able to return for the Post-Implant 6-Month Device Follow-Up Visit

Exclusion Criteria:

* Are ≤19 years of age (due to specifications outlined in cognitive function test requirements)
* Are ≥90 years of age (due to specifications outlined in cognitive function test requirements)
* Are pregnant at time of enrolment
* Is participating in an investigational drug investigation
* Be experiencing a condition at the time of data collection which affects mental capacity (lack capacitiy), such as dementia, Alzheimer's, psychosis, schizophrenia (excluding depression and anxiety).
* Recent Cerebral Vascular Event (CVE) which may have affected cognitive function
* Heavy substance abuse, drugs or alcohol

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients (left ventricular ejection fraction (LVEF) <35%) receiving an Cardiac Implantable Electronic Device (CIED), including Cardiac Resynchronisation Therapy (CRT), an Implantable Cardioverter Defibrillator (ICD) or a Permanent Pacemaker (PPM).
Sampling Method: Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2024-01-14 (Estimated); Study Completion 2024-01-14 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function at 6 months post-implant | 6 months
  Measured by the use of a 5-stage cognitive battery test

SECONDARY OUTCOMES:
Change in left ventricular ejection fraction (LVEF) at 6 months | 6 months
  Measured by transthoracic echocardiogram (TTE)
Change in N-terminal pro-B-type natriuretic peptide (NT-proBNP) Test at 6 months | 6 months
  Measured by a NT-proBNP blood test.
Change in New York Heart Association (NYHA) Functional Classification | 6 months
  Measured via standardised assessment for all participants

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Ford, BSc (Hons), Principal Investigator — Royal Cornwall Hospital NHS Trust
Locations (1):
- Royal Cornwall Hospital NHS Trust, Truro, Cornwall, United Kingdom

IPD SHARING:
Plan to Share IPD: No